CLINICAL TRIAL: NCT04067908
Title: Study of New Biomarkers Associated With the Risk of Premature Delivery During Spontaneous Work With Intact Membranes Before 37 Weeks of Amenorrhea.
Brief Title: New Biomarkers Associated With the Risk of Premature Delivery.
Acronym: PROTEOMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2010/19
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Premature Delivery
Keywords: Biological markers
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- woman giving birth prematurely (Experimental): Proteome: by liquid chromatography coupled with tandem mass spectrometry. Fibronectin: by vaginal sampling. Ultrasound of the cervix. Cytokines: ELISA kit of a panel of several cytokines.
  Interventions: Other: 2 tubes of 5ml during the blood collection and 2 swabs during vaginal sampling

INTERVENTIONS:
Other: 2 tubes of 5ml during the blood collection and 2 swabs during vaginal sampling — The samples taken during this study are taken at the same time as those taken in routine during the diagnosis of threat of premature labor. There are added 2 tubes of 5ml during the blood collection and 2 swabs during vaginal sampling.

SUMMARY:
Despite the progress made in the organization of care and neonatal care, prematurity remains the main cause of morbidity and perinatal mortality.

This study aims to estimate the prognostic value of new biomarkers (proteomic markers) on the occurrence of preterm birth.

DETAILED DESCRIPTION:
Despite the progress made in the organization of care and neonatal care, prematurity remains the main cause of morbidity and perinatal mortality. With 7.2% of premature deliveries in France, threat of premature labor remains the leading cause of maternal transfer and hospitalization. In terms of mortality, morbidity and cost, the fight against prematurity remains a national priority in terms of public health.

The diagnosis of threat of premature labor at high risk of preterm labor is difficult and clinical and laboratory criteria often remain insufficient. Measurement of the cervix by endovaginal ultrasound lacks sensitivity and specificity. Among the biological criteria, only fibronectin, which has a good negative predictive value, is used in current practice. Despite the use of these two prognostic criteria, only 40% of hospitalized patients will give birth prematurely.

Recent advances in proteomics allow us to study complex proteomes and compare them. Preliminary studies already carried out have revealed families of proteins expressed differently in situations of work or premature delivery. We therefore hypothesize that the study of a woman's vaginal proteome with threat of premature labor may reveal new markers of preterm labor. These markers could help the clinician in its therapeutic management and thus reduce hospitalizations, better target patients requiring tocolytic treatment and optimize the use of corticosteroids. In addition, variations in the proteome may help to understand the physiopathological mechanisms of premature delivery, which are necessary for the development of effective therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 18 years of age
* Term from 22 to 33 and 6 amenorrhea weeks
* Single or twin pregnancy
* Emergency consultant, in participating centers, for a threat of premature labor defined by:

Uterine contractions greater than or equal to 3 in 30 minutes Clinical modification of the cervix Ultrasound collar less than 25 mm

* Free, informed and written consent, dated and signed by the patient and the investigator before any investigation required by the research.
* Patient affiliated to a Social Security scheme.

Exclusion Criteria:

* Premature rupture of membranes
* Placenta previa
* Vaginal haemorrhage at the time of sampling
* Uterine malformation
* Strapping, open bite
* History of strapping and or open bite
* Conization
* Fetal malformation
* Associated vasorenal pathology
* Sexual intercourse less than 24h
* Gynecological examination less than 48h
* Vaginal treatment in progress
* Polyhydramnios
* Transfused-transfused syndrome
* Twin Anemia Polycythemia syndrome
* Fetoscopy during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman during childbirth
Enrollment: 182 (Actual)
Dates: Start 2011-06-07 (Actual); Primary Completion 2013-12-28 (Actual); Study Completion 2013-12-28 (Actual)

PRIMARY OUTCOMES:
Premature delivery yes/no | Premature delivery before 33 amenorrhea weeks + 6 days
  Premature labor is defined as a pregnancy duration of less than 37 weeks. For this study, cases of interest are : premature labor before 33 amenorrhea weeks + 6 days.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique DALLAY, Pr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No